CLINICAL TRIAL: NCT03539770
Title: Lung Regeneration After Posterior Spinal Fusion for Adolescent Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: CIN_LungRegenAIS_001
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Scoliosis Idiopathic Adolescent
Keywords: Lung Development; Lung Regeneration; Hyperpolarized Helium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AIS: Adolescent idiopathic scoliosis subjects undergoing posterior spinal fusion.
  Interventions: Procedure: Posterior spinal fusion
- Control: Children without scoliosis

INTERVENTIONS:
Procedure: Posterior spinal fusion — Surgical procedure that involves placement of spinal rods to correct spinal curvature
  Groups: AIS

SUMMARY:
Adolescent Idiopathic Scoliosis (AIS) is a curvature of the spine that occurs in 1-2% of otherwise healthy children, and requires corrective surgery, posterior spinal fusion (PSF) in ~10% of cases. Some studies suggest that pulmonary function is reduced in AIS and that PSF improves pulmonary function. The lung is composed of a large number of branching airways that terminate in gas exchanging units called alveoli, and the number and structure of these alveoli are partially dependent upon lung volume and the forces to which they are exposed--two factors predicted to be altered in AIS. This study uses MRI imaging of inhaled helium to quantify alveolar structure in children with and without AIS before and one-year after PSF. The goals of the study are to determine if alveolar architecture or number are altered in AIS and whether PSF impacts these same measures.

DETAILED DESCRIPTION:
After obtaining informed consent, subjects are trained in a breath holding technique that permits obtaining reproducible proton and hyperpolarized helium (HHE) lung images. 3-Helium is obtained from a vendor and hyperpolarized using an optical spin transfer device (FDA Investigational New Drug (IND) 122,670) and administered through a valved inhalation device while in the MRI scanner. Images are obtained during an ~15 second inspiratory breath hold. Proton MRI images are similarly obtained during a breath hold with room air using an ultrashort echo time sequence. From these MRI images, lung volumes, alveolar sizes, and estimated alveolar numbers are derived. Subjects are reimaged at 1 year to evaluate changes in these parameters during normal lung growth (controls) or after PSF (AIS subjects).

ELIGIBILITY:
Inclusion Criteria:

1. Be diagnosed with AIS.
2. Have a Cobb Angle > 50°.
3. Be recommended for PSF.
4. Be between the ages of 8 and 21 years old (inclusive) at the time of surgery.
5. Be able to perform the required 10 second inspiratory hold and remain lying still for that time period without the need for sedative medication (as assessed at time of enrollment).
6. Have a primary caregiver who agrees to attend all required points of contact for this study (if under the age of 18).

Exclusion Criteria:

1. Have had a previous spinal surgery.
2. Have other planned major surgeries during the study period.

   a. Minor surgeries such as G-tube revisions or dental procedures are permissible.
3. Have or had a history of any chronic lung disease apart from restrictive lung disease from scoliosis (e.g.

   cystic fibrosis, bronchopulmonary dysplasia, asthma, etc.).
4. Have a personal history of smoking
5. Require any supplemental oxygen at baseline. Home Biphasic Positive Airway Pressure (BiPAP) or Continuous Positive Airway Pressure (CPAP) is acceptable provided the participant can perform the required breath holds without these devices.
6. Have been born at <35 weeks gestational age.
7. Received mechanical ventilation in the first year of life.
8. Have a room air oxygen saturation of less than 95%.
9. Have any implanted metal device or hardware (apart from future orthopaedic hardware).
10. Be likely to move out of the Cincinnati area before the one year follow-up appointment.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Healthy control and otherwise healthy AIS children and young adults
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Alveolar Size | Before posterior spinal fusion and one year after
  Calculated mean linear intercept as determined by diffusion measurements in HHe MRI

SECONDARY OUTCOMES:
Change in Lung Volume | Before posterior spinal fusion and one year after
  Measured right and left lung volumes as measured by proton MRI
Change in Alveolar Number | Before posterior spinal fusion and one year after
  Estimated number of alveoli in right and left lung as calculated from alveolar size and lung volume measures
Altered Alveolar Size in AIS | 1 day
  Determine differences in mean linear intercept (MLI) as determined by HHe diffusion measurements in AIS vs control and AIS right vs left lung
Differences in Lung Volume in AIS | 1 day
  Determine differences in lung volume as determined by proton MRI in AIS vs control and AIS right vs left lung
Differences in Alveolar Number in AIS | 1 day
  Determine differences in estimated alveolar number as calculated using MLI and lung volume measures in AIS vs control and AIS right vs left lung

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
We would be willing to share individual participant data with researchers who request the data.

REFERENCES:
- [Derived] Thomen RP, Woods JC, Sturm PF, Jain V, Walkup LL, Higano NS, Quirk JD, Varisco BM. Lung microstructure in adolescent idiopathic scoliosis before and after posterior spinal fusion. PLoS One. 2020 Oct 8;15(10):e0240265. doi: 10.1371/journal.pone.0240265. eCollection 2020. PMID 33031412